CLINICAL TRIAL: NCT04443816
Title: Advanced Geriatric Evaluation in Predicting Health Related Quality of Life in Patients With Colorectal Cancer
Brief Title: Advanced Geriatric Evaluation and Quality of Life in Colorectal Cancer Surgery
Acronym: AGE CRC
Status: Completed | Type: Observational
Sponsor: St. Antonius Hospital (Other)
Responsible Party: Principal Investigator, dr. P. Noordzij, Principal Investigator, St. Antonius Hospital
Other Study IDs: NL6152310017
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) disproportionately affects patients aged 70 years and older. Surgery is the main treatment modality for CRC, but is associated with increased risk of postoperative morbidity, disability and loss of health related quality of life (HRQL).Frailty is an age related state of functional decline and considered to be an important risk factor for adverse outcome in geriatric oncology.Risk models for adverse outcome may be used for treatment decisions in the elderly, but are often not designed to predict patient related outcome measures and do not include frailty characteristics.

DETAILED DESCRIPTION:
Multicentre, prospective, observational cohort study with a follow up time of one year. After initial diagnosis of CRC subjects will be screened for frailty using validated questionnaires, physical tests and non-invasive measurements. Frailty characteristics and HRQL are determined by Geriatric 8 (G8), Hospital Anxiety and Depression Scale(HADS), Euroqol- 5 dimensional (EQ-5D), Lawton Instrumental Activity of Daily Living scale(IADL), Mini Nutrition Assessment (MNA), 6 Item Cognitive Impairment Test (6-CIT), Identification of Seniors At Risk - Hospitalized Patients(ISAR-HP) and the EORTC-QLQ-C30/CR29 (HRQL in CRC patients). Physical tests include the Timed to Get Up (TUG) test and the hand grip strength test. Furthermore, the non-invasive measurements consist of a sarcopenia analysis using an existing CT/MRI scan and measurement of Advanced Glycation Endproducts (AGE reader).

Additional patients characteristics including medication use, medical history, tumor characteristics, neoadjuvant therapy and laboratory results of preoperative routine blood sampling will be collected. At three, six and twelve months after diagnosis, EORTC QLQ-C30/EORTC QLQ-CR29 and EQ-5D questionnaires are used to determine HRQL and disability free survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years
* Histologically proven non-metastatic colorectal cancer
* Signed informed consent

Exclusion Criteria:

* - Emergency surgical procedures
* Insufficient understanding of the Dutch language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: aged ≥ 70 years with a new diagnosis of non-metastatic CRC
Sampling Method: Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-06 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Loss of health related quality of life (HRQL) | 12 months
  Change in EORTC QLQ-C30

SECONDARY OUTCOMES:
Loss of health related quality of life (HRQL) | 3 months
  Change in EORTC QLQ-C30
Postoperative complications | 30 days
  Complication after surgery
Disability | 12 months
  EQ-5D

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Meander medical center, Amersfoort
  - Tergooi hospital, Hilversum
  - St Antonius Hospital, Nieuwegein
  - Rivierenland ziekenhuis, Tiel
  - Diakonessenhuis, Utrecht
  - UMCU, Utrecht

REFERENCES:
- [Derived] van der Vlies E, Vernooij LM, Hamaker ME, van der Velden AMT, Smits M, Intven MPW, van Dodewaard JM, Takkenberg M, Vink GR, Smits AB, Bos WJW, van Dongen EPA, Los M, Noordzij PG. Frailty and health related quality of life three months after non-metastatic colorectal cancer diagnosis in older patients: A multi-centre prospective observational study. J Geriatr Oncol. 2022 Jan;13(1):74-81. doi: 10.1016/j.jgo.2021.08.005. Epub 2021 Aug 24. PMID 34446378